CLINICAL TRIAL: NCT06770868
Title: A Novel Alloplastic Patient Specific Temporalis Tendon Enthesis for Mandibular Resection with Coronoidectomy
Brief Title: A Novel Alloplastic Patient Specific Temporalis Tendon Enthesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0118-21/24
Record Dates: First submitted 2024-12-21; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Mandibular Resection
Keywords: mandibular resection; coronoid; computer assisted; computer-aided design,; computer-aided manufacturing

STUDY DESIGN:
Intervention Model Description: mandibular resection with coronoidectomy managed with patient specific reconstruction plate with custom made temporalis tendon enthesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient specific reconstruction plate for patients suffering from mandibular segmental defects (Experimental): Patients with mandibular segmental defect including coronoidectomy managed with patient specific reconstruction plate with custom made temporalis tendon enthesis
  Interventions: Device: Patient specific reconstruction plate for patients suffering from mandibular segmental defects

INTERVENTIONS:
Device: Patient specific reconstruction plate for patients suffering from mandibular segmental defects — Patients with mandibular segmental defect including coronoidectomy managed with patient specific reconstruction plate with custom made temporalis tendon enthesis

SUMMARY:
Mandibular reconstruction of segmental defects is an arduous surgical procedure that requires an utmost degree of surgical fidelity. Whether primary bone reconstruction is feasible or not, alloplastic bridging between the remaining bone stumps is mandatory to achieve functional, aesthetic, and symmetrical demands of the lower third of the face. Mandibular reconstructive surgery should be directed toward the maintains of the normal orthognathic centric condylar position, mandibular kinematics, and muscles of mastication function. Mandibular resection with coronoid removal cause imbalance in the attachment of one of the large muscles of mastication, the temporalis muscle. The use of computer-aided surgery allowed the creation of custom made fixation plates with a plethora of advantages over the conventional plates.

the study aims to introduce a novel plate design, which creates an enthsis for the reattachment of the temporalis muscle tendon.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular lesion that require segmental resection.
* Patients required coronoid processes resection within the safety margin of the lesion.
* Brown Class I cases with preservation of the condyle process and no need for alloplastic TMJ replacement.
* Complaisant patient that is able to complete at least 1 year follow up.

Exclusion Criteria:

* Composite mandibular defect.
* Malignant lesions that required postoperative adjunctive therapies (CT or RT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Mandibular Kinematics assessment | 6 months
  range of mandibular excursions were recorded preoperatively (T0) and at 1-postopertive week (T1), 1-postoperative month (T2), 4-postoperative month (T3), 6- postoperative month (T4).

SECONDARY OUTCOMES:
Postoperative temporalis muscle activity | 6 months
  surface-Electromyogram (sEMG) was used by the patients during their maximum voluntary clenching by placement of two channels on the bilateral temporalis muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP
Access Criteria: to any one who required them after deidentification